CLINICAL TRIAL: NCT03196752
Title: Utility of the Laryngeal Handshake Method for Identifying the Cricothyroid Membrane
Brief Title: Laryngeal Handshake for Identifying the Cricothyroid Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ho Geol Ryu, Assistant professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1704-035-844
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Emergent Cricothyrodotomy
Keywords: cricothyroid membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Only arm (Experimental): Patient's cricoid membrane is identified using both laryngeal handshake method and simple palpation
  Interventions: Procedure: laryngeal handshake; Other: simple palpation

INTERVENTIONS:
Procedure: laryngeal handshake — palpate for the cricothyroid membrane using the laryngeal handshake technique
Other: simple palpation — conventional

SUMMARY:
The cricothyroid membrane is the most common position that the invasive airway secure is performed, but it is not easy to identify the cricothyroid membrane by tactile perception. Although it is recommended to use the laryngeal handshake method for identifying the cricothyroid membrane in difficult airway society 2015 guidelines for management of unanticipated difficult intubation in adults, there is only suggestion without clinical data about how much the laryngeal handshake method improves the accuracy of identification of the cricothyroid membrane So we made the hypothesis that the cricothyroid membrane is identified more correctly when the laryngeal handshake method is used than when that method is not used. And we try to find out whether there is actual difference about identification of the cricothyroid membrane between using the laryngeal handshake method and not using that method. By identifying the difference between them, we are going to support the recommendation of guidelines and make the evidence for educating the doctors who have any possibility to perform the criocthyroidotomy to use the laryngeal handshake method skillfully in the 'cannot intubate, cannot oxygenate' situation.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent nose or ear surgery in Seoul National University Hospital and Seoul Metropolitan Government Seoul National University Boramae Medical Center

Exclusion Criteria:

* those whose ASA class was over 3, those who rejected to participate study or had impaired capacity to agree, those who was going to undergo neck surgery, those who had anatomical anomaly or skin lesion at neck, and those who were pregnant were excluded.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
accuracy of cricothyroid membrane identification | Baseline
  accuracy between conventional identification of the cricothyroid membrane and the laryngeal handshake method

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul, Agree
  - Boramae Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oh H, Yoon S, Seo M, Oh E, Yoon H, Lee H, Lee J, Ryu HG. Utility of the laryngeal handshake method for identifying the cricothyroid membrane. Acta Anaesthesiol Scand. 2018 Oct;62(9):1223-1228. doi: 10.1111/aas.13169. Epub 2018 Jun 21. PMID 29926892